CLINICAL TRIAL: NCT04305340
Title: Bio-signal Telemonitoring Using Electronic Textiles in a Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aamir Jeewa (Other)
Collaborators: Toronto Rehabilitation Institute (Other)
Responsible Party: Sponsor-Investigator, Aamir Jeewa, Staff Cardiologist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTO 1891
Record Dates: First submitted 2019-11-29; First posted 2020-03-12 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Pediatric; Smart Device; Remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SKIIN Textile Device in children with healthy hearts (Experimental): The Myant SKIIN Device will be worn by study participants while they lay down, sit, stand, exercise and cool-down.
  Interventions: Device: Myant SKIIN Device
- SKIIN Textile Device in children with heart failure (Experimental): The Myant SKIIN Device will be worn by study participants while they lay down, sit, stand, exercise and cool-down
  Interventions: Device: Myant SKIIN Device

INTERVENTIONS:
Device: Myant SKIIN Device — 1. Supine position: Participant lays on a bed on their back for 5 minutes
  2. Sitting position: Participant sits on a chair for 5 minutes
  3. Standing position: Participant stands for 5 minutes.
  4. Exercise measurement: treadmill exercise test - the protocol entails increases of 0.5 mph every minute with zero change in the incline. Starting point would 1.5 mph. The test will be interrupted if the target heart rate of 190 beats per minute is reached or if symptoms and/or arrhythmias and ST depression would be observed. Patient will be monitor during recovery for 5 minutes.
  5. Cool-down: Participants cool-down for 5 minutes

SUMMARY:
There is a need for developing reliable and convenient technologies for telemonitoring of physiological signals such as respiration, cardiac function, and activity level in children and especially for those with heart disease. Changing symptomatology causes heart failure patients to seek medical attention in order to be assessed and potentially have medication adjusted or additional testing being undertaken. These frequent clinical encounters affect the quality of life of these children and their parents, as well as being costly for the health care system. A textile based technology for telemonitoring application that is comfortable and accurate in its data collection can help to provide real time information on physiologic parameters. The primary research objective is to determine the feasibility and validity of a textile-enabled sensor system in measuring physiologic variables, or "biological signals", related to cardiopulmonary function in children. The study will include 10 patients with heart failure, and 10 healthy controls.

ELIGIBILITY:
Inclusion Criteria

1. Healthy children participants (i.e. without CHD or HF) aged between 10 to 18 years with normal electrocardiograms and normal echocardiograms (i.e. screens for familial cardiomyopathy).

   OR
2. Patients aged between 10 and 18 years with diagnosed congenital heart disease or cardiomyopathies referred to pediatric cardiology ambulatory clinic at SickKids.

Exclusion Criteria

1. In-hospital patients.
2. Patients too ill to participate or perform any activity.
3. Patients with Fontan/single ventricle physiology circulation.
4. Children who are less than 6 months post op from a cardiac surgery as they will have concerns from an activity and wound care standpoint.
5. Participants with known allergies to adhesives (as reported by family).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Validate the heart rate measurements obtained using the SKIIN Textile in children with and without heart disease. | 40 minutes
  Validate the heart rate measurements obtained using the SKIIN Textile in children with and without heart disease compared to the measurements obtained by the Grael 4K PSG
Validate the respiratory rate measurements obtained using the SKIIN Textile in children with and without heart disease. | 40 minutes
  Validate the respiratory rate measurements obtained using the SKIIN Textile in children with and without heart disease compared to the measurements obtained by the Grael 4K PSG.
Validate the pulse oximetry measurements obtained using the SKIIN Textile in children with and without heart disease. | 40 minutes
  Validate the pulse oximetry measurements obtained using the SKIIN Textile in children with and without heart disease compared to the measurements obtained by the Nonin, WristOx2TM, Model 3150, Wrist-worn Pulse Oximeter

SECONDARY OUTCOMES:
To extract and analyze temperature data obtained using the SKIIN Textile in children with | 40 minutes
  To extract and analyze temperature data obtained using the SKIIN Textile in children with

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Jeewa, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No